CLINICAL TRIAL: NCT00622336
Title: Open-Label, Single-Arm Study of the Safety and Efficacy of CC-5013 Monotherapy for Subjects With Multiple Myeloma: A Companion Study for Studies THAL-MM-003, CC-5013-MM-009, and CC-5013-MM-010
Brief Title: A Companion Study for Studies THAL-MM-003, CC-5013-MM-009, and CC-5013-MM-010 for Subjects With Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-5013-MM-012; 2004-002102-30 (EudraCT Number)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Revlimid
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide 25mg (CC-5013) (Experimental): Oral 25mg daily on Days 1-21 every 28 days
  Interventions: Drug: CC-5013; Drug: Lenalidomide

INTERVENTIONS:
Drug: CC-5013 — Oral 25mg daily on Days 1-21 every 28 days.
  Other Names: Revlimid; lenalidomide
Drug: Lenalidomide — Oral Lenalidomide 25mg daily on Days 1-21 every 28 days.
  Other Names: Revlimid; CC-5013

SUMMARY:
The study evaluated the safety of Lenalidomide monotherapy in participants with advanced multiple myeloma who had discontinued treatment with combination thalidomide plus high-dose dexamethasone or high-dose dexamethasone alone in studies Thal-MM-003, CC-5013-MM-009 and CC-5013-MM-010 due to the development of documented disease progression or the inability to tolerate the lowest dosing regimen per previous protocol of thalidomide and/or high-dose dexamethasone without grade 3 or 4 toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Age ≥ 18 years at time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements
* Participants with multiple myeloma and were enrolled in either THAL-MM-003, CC-5013-MM-009, or CC-5013-MM-010 and discontinued study therapy with thalidomide and high-dose dexamethasone or high-dose dexamethasone alone due to:

documented disease progression OR inability to tolerate the lowest dosing regimen allowed on previous protocol without a grade 3 or 4 toxicity.

* Eastern Cooperative Oncology Group (ECOG) performance status score 0,1,2
* Recovery from thalidomide or dexamethasone-related toxicity to ≤ grade 2 (NCI CTC)
* Females of child-bearing potential (FCBP) must agree to using two methods of contraception

Exclusion Criteria:

* Prior development of a ≥ grade 2 allergic reaction/hypersensitivity or prior development of a grade ≥ 3 rash or desquamation while taking thalidomide National Cancer Institute Common toxicity Criteria (NCI CTC)
* Use of any standard/experimental anti-myeloma therapy within 28 days of randomization or use of any experimental non-drug therapy within 56 days of initiation of drug treatment
* Any serious medical condition, laboratory abnormality, or psychiatric illness that will prevent the participant from signing the informed consent form or that will place the participant at an unacceptable risk for toxicity if he/she participates in the study.
* Pregnant or lactating females.
* Prior therapy with CC-5013; prior history of malignancies, other than multiple myeloma (except basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast), unless subject has been free of disease for ≥ 5 years
* More than 4 months has elapsed since the last dose of study drug was administered on study Tal MM-003, CC-5013-MM-009, CC-5013-MM-010
* Absolute neutrophil count (ANC) <1,000cells/mm^3 (1.0 X 10^9/L)
* Platelet count <75,000/mm^3 (30 X 10^9/L) for those with <50% if the bone marrow nucleated cells re plasma cells; Platelet count <30,000/mm^3 (30 X 10^9/L) for those with <50% if the bone marrow nucleated cells re plasma cells
* Serum creatinine >2.5mg/dL; serum SGOT/AST or SGPT/ALT x upper limits of normal (ULN)
* Serum total bilirubin >2.0mg/d/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2003-04-01 (Actual); Primary Completion 2013-11-25 (Actual); Study Completion 2013-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Knight, MD, Study Director — Celgene Corporation
Locations (7):
- Russia (4):
  - Republican Clinical Hospital #1, Izhevsk
  - Nizhny Novgorod Clinical Hospital n.a.Semashko, Nizhny Novgorod
  - Novosibirsk State Regional Clinical, Novosibirsk
  - Samara Regional Clinical Hospital, Samara
- Ukraine (3):
  - Kharkov Postgraduate Medical Academy Kharkov Regional Clinical, Kharkiv
  - Institute of Hematology and Transfusiology of the UAMS Department of blood diseases, Kiev
  - Odessa Regional Clinical Hospital, Odesa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an international, open-label single arm study of oral lenalidomide in participants with multiple myeloma who had previously received high dose dexamethasone alone or in combination with thalidomide in the study NCT 00057564, or previously received high dose dexamethasone alone in studies NCT 00056160 and NCT 00424047.
Pre-assignment Details: To be eligible participants must have developed disease progression or were unable to tolerate the lowest dosing regimen of thalidomide and/or high-dose dexamethasone without Grade 3 or 4 toxicity
Groups:
- Lenalidomide 25mg: Lenalidomide 25mg by mouth (PO) daily on Days 1 to 21 in each 28 day cycle
Period: Treatment Phase
Arm/Group | Lenalidomide 25mg
Started | 330
Safety Population | 330
Completed | 21 (Completed = those who completed the treatment phase and were ongoing in the extension study)
Not Completed | 309
Not completed — Progression of Disease | 181
Not completed — Adverse Event | 46
Not completed — Other | 40
Not completed — Death | 14
Not completed — Lack of therapeutic effect | 13
Not completed — Withdrawal by Subject | 13
Not completed — Lost to Follow-up | 2
Period: Extension Phase
Arm/Group | Lenalidomide 25mg
Started | 21
Completed | 0
Not Completed | 21
Not completed — Adverse Event | 2
Not completed — Progressive Disease | 6
Not completed — Lack of therapeutic effect | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide 25mg (CC-5013)
Number analyzed (Participants) | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (9.43)
Age, Customized [Number; unit: participants]
  > 65 years | 136
  ≤ 65 years | 194
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 193
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian/Pacific Islander | 2
  Black or African American | 14
  White | 309
  Hispanic | 5
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a patient's disease is progressing, assess how the disease affects the daily living activities of the patient and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = Fully Active | 95
    1 = Restricted Activity | 178
    2 = Ambulatory; not able to work | 44
    3 = Limited Self Care | 1
    4 = Completely Disabled | 0
    Missing= Unspecified | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AE) During the Treatment Phase
Description: An AE is any sign, symptom, illness, or diagnosis (either observed or volunteered) that appears or worsens during the course of the study Serious adverse event (SAE) = any AE which results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect; constitutes an important medical event. A treatment emergent AE is defined as any AE occurring or worsening on or after the first dose of study drug and within 30 days after the last dose of study drug. Safety and severity was assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 2.0; Severity of AEs were graded (including second primary malignancies) as Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe; Grade 4- Life-threatening; Grade 5-Fatal;
Time Frame: Until data cut-off of 22 Oct 2009; AEs/SAEs were recorded from informed consent to 30 days post treatment discontinuation visit. Maximum exposure to Lenalidomide treatment was 1260 days.
Population: The safety population included participants enrolled in the study and had received at least one dose of lenalidomide.
Measure: Number; unit: participants
Arm/Group | Lenalidomide 25mg (CC-5013)
Number analyzed (Participants) | 330
participants
  Adverse Event (AE) | 327
  Adverse Event related to study drug | 268
  Adverse Event NCI CTC (Version2.0) Grade 3 or 4 | 256
  Serious Adverse Event (SAE) | 177
  AE leading to discontinuation of study drug | 52
  AE leading to dose reduction/interruption | 210

2. Secondary Outcome: Time to Progression
Description: Time to progression based on the myeloma response determination criteria developed by Bladé et al 1998 and is defined as the time from registration to the first documented progression. The progressive disease criteria included increasing monoclonal paraprotein levels, bone marrow findings, worsening lytic bone disease, progressively enlarging extramedullary plasmacytomas, or hypercalcemia.
Time Frame: Up to 70 months
Population: Time to progression not analyzed per the sponsors decision.
Arm/Group | Lenalidomide 25mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Myeloma Response Rate
Description: Myeloma response determination criteria developed by Bladé et al 1998. Complete Response (CR):Disappearance of monoclonal paraprotein. Remission Response (RR):75-99% reduction in monoclonal paraprotein/90-99% reduction in 24-hr urinary light chain excretion. Partial Response (PR):50-74% reduction in monoclonal paraprotein/50-89% reduction in 24-hr urinary light chain excretion. Stable Disease (SD):Criteria for PR or PD not met. Plateau Phase:If PR, stable monoclonal paraprotein (within 25% above or below nadir)/stable soft tissue plasmacytomas. Progressive Disease (PD):Disease worsens.
Time Frame: Up to 70 months
Population: Myeloma Response Rate not analyzed per the sponsors decision.
Arm/Group | Lenalidomide 25mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Duration of Response
Description: Duration of response based on the Myeloma response determination criteria developed by Bladé et al 1998 and defined as time from the initial documented response (partial response or better) to confirmed disease progression, based on International Myeloma Working Group (IMWG) criteria.
Time Frame: Up to 70 months
Population: Duration of response not analyzed per the sponsors decision.
Arm/Group | Lenalidomide 25mg
Number analyzed (Participants) | 0

5. Primary Outcome: Number of Participants With Adverse Events (AE) During the Extension Phase
Description: as for outcome 1
Time Frame: From 22 Oct 2009 to November 2013; AEs/SAEs were recorded from informed consent to 30 days post treatment discontinuation visit.
Population: Included participants who were enrolled in the extension phase. The safety population included participants enrolled in the study and had received at least one dose of lenalidomide.
Measure: Number; unit: participants
Arm/Group | Lenalidomide 25mg (CC-5013)
Number analyzed (Participants) | 21
participants
  ≥ 1 Adverse Event (AE) | 13
  Adverse Event related to study drug | 1
  Adverse Event NCI CTC (Version2.0) Grade 3 or 4 | 5
  ≥ 1 Serious Adverse Event (SAE) | 5
  ≥ 1 AE leading to discontinuation of study drug | 1
  ≥ 1 AE leading to dose reduction/interruption | 3

ADVERSE EVENTS:
Time Frame: From first dose of study drug through to 30 days after the last dose, until the data cut-off date of 11 November 2013. Maximum time on Lenalidomide treatment was 1260 days.
Groups:
- Lenalidomide (Treatment Phase) Up to Data Cut-off 22 Oct 2009; Lenalidomide ( ExtensionPhase) 22 Oct 2009 to 11 November 2013: Lenalidomide 25mg by mouth (PO) daily on Days 1 to 21 in each 28 day cycle
Arm/Group | Lenalidomide (Treatment Phase) Up to Data Cut-off 22 Oct 2009 | Lenalidomide ( ExtensionPhase) 22 Oct 2009 to 11 November 2013
Serious Adverse Events (participants affected / at risk) | 177/330 | 5/21
Other Adverse Events (participants affected / at risk) | 0/330 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Treatment Phase) Up to Data Cut-off 22 Oct 2009 (N=330) | Lenalidomide ( ExtensionPhase) 22 Oct 2009 to 11 November 2013 (N=21)
Pneumonia NOS (Infections and infestations) | 38 | 2
Respiratory tract infection NOS (Infections and infestations) | 6 | 0
Lobar pneumonia NOS (Infections and infestations) | 4 | 0
Sepsis NOS (Infections and infestations) | 4 | 0
Bacteraemia (Infections and infestations) | 3 | 0
Bronchitis acute NOS (Infections and infestations) | 3 | 0
Bronchopneumonia NOS (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Lung infection NOS (Infections and infestations) | 2 | 0
Pyelonephritis NOS (Infections and infestations) | 2 | 0
Abscess NOS (Infections and infestations) | 1 | 0
Arthritis infective NOS (Infections and infestations) | 1 | 0
Bronchitis chronic NOS (Infections and infestations) | 1 | 0
Candida pneumonia (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Haemophilus sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection NOS (Infections and infestations) | 1 | 0
Obstructive chronic bronchitis with acute exacerbation (Infections and infestations) | 1 | 0
Osteomyelitis NOS (Infections and infestations) | 1 | 0
Osteomyelitis chronic NOS (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pyelonephritis chronic NOS (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Urinary tract infection NOS (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Varicella (Infections and infestations) | 1 | 0
Viral infection NOS (Infections and infestations) | 1 | 0
Anaemia NOS (Blood and lymphatic system disorders) | 11 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 0
Leukopenia NOS (Blood and lymphatic system disorders) | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 4 | 0
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 14 | 0
Asthenia (General disorders) | 7 | 0
Multi-organ failure (General disorders) | 2 | 0
Disease progression NOS (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 1
Injection site cellulitis (General disorders) | 1 | 0
Lethargy (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Gastroenteritis NOS (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Diarrhoea NOS (Gastrointestinal disorders) | 3 | 1
Abdominal pain NOS (Gastrointestinal disorders) | 2 | 0
Oesophagitis NOS (Gastrointestinal disorders) | 2 | 0
Periproctitis (Gastrointestinal disorders) | 2 | 0
Appendicitis (Gastrointestinal disorders) | 1 | 0
Diverticulitis NOS (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastritis NOS (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain NOS (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia NOS (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction NOS (Gastrointestinal disorders) | 1 | 0
Umbilical hernia NOS (Gastrointestinal disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Jaw osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Bronchitis NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive airways disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary thrombosis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 0
Cardiac failure NOS (Cardiac disorders) | 3 | 0
Pulmonary oedema NOS (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Coronary artery disease NOS (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 0
Subdural haematoma (Nervous system disorders) | 2 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebrovascular disorder NOS (Nervous system disorders) | 1 | 0
Dementia NOS (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Metabolic encephalopathy NOS (Nervous system disorders) | 1 | 0
Phantom pain (Nervous system disorders) | 1 | 0
Radiculitis brachial (Nervous system disorders) | 1 | 0
Spinal cord compression NOS (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain neoplasm NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carcinoid tumour NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Craniopharyngioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Light chain disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal adenocarcinoma NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 6 | 0
Renal failure NOS (Renal and urinary disorders) | 4 | 0
Calculus urinary (Renal and urinary disorders) | 2 | 0
Nephropathy NOS (Renal and urinary disorders) | 2 | 0
Renal failure acute or chronic (Renal and urinary disorders) | 2 | 1
Azotaemia (Renal and urinary disorders) | 1 | 0
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0
Accident NOS 1 ( 0.3) (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Intracranial injury NOS (Injury, poisoning and procedural complications) | 1 | 0
Perirenal haematoma (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture NOS (Injury, poisoning and procedural complications) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus NOS (Metabolism and nutrition disorders) | 2 | 0
Hyperproteinaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 0
Hypotension NOS (Vascular disorders) | 2 | 0
Aortic thrombosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 0
Agitation (Psychiatric disorders) | 1 | 0
Conversion disorder (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Cholecystitis acute NOS (Hepatobiliary disorders) | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis NOS (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Liver function tests NOS abnormal (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Rash NOS (Skin and subcutaneous tissue disorders) | 2 | 0
Dermatitis medicamentosa (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia of Malignant Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (Treatment Phase) Up to Data Cut-off 22 Oct 2009 (N=330) | Lenalidomide ( ExtensionPhase) 22 Oct 2009 to 11 November 2013 (N=21)
Anaemia NOS (Blood and lymphatic system disorders) | 0 | 2
Asthenia (General disorders) | 0 | 3
Headache (Nervous system disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator has the right to publish and/or present study data after multicentric publication or one year has elapsed until completion this multicentric study provided that he/she (i) furnishes the sponsor a copy of any proposed publication or presentation before its submission, (ii) deletes any sponsor's confidential data as pointed out by sponsor, and (iii) delays any submission for generally up to ninety (90) days to permit the preparation and filing of intellectual property applications.